CLINICAL TRIAL: NCT03986697
Title: In Patients Taking Protease Inhibitors Does Switching to a Bictegravir, Tenofovir Alafenamide and Emtricitabine Combination, Reduce Cardiovascular Risk: an Open-label, Randomised, Serial CT Pilot Study
Brief Title: How Does Antiretroviral Therapy Affect Coronary Atherosclerosis: a Serial CT Study
Acronym: HART CT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID19 emergency. No patients randomised
Sponsor: University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UoL001362; 2017-005033-22 (EudraCT Number)
Record Dates: First submitted 2019-05-30; First posted 2019-06-14 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2019-09

CONDITIONS: Coronary Artery Disease; Hiv
Keywords: HIV; Coronary Artery Disease; Atherosclerosis; Antiretroviral therapy; Computed tomography
MeSH Terms: conditions — Coronary Artery Disease; Acquired Immunodeficiency Syndrome; Atherosclerosis | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bictarvy (Active Comparator): Intervention group: those randomised to switch antiretroviral therapy to Bictegravir, Emtricitabine and Tenofovir Alafenamide fixed dose combination.
  Interventions: Drug: Biktarvy
- Usual therapy (No Intervention): Control group: those randomised to continue their usual antiretroviral regime

INTERVENTIONS:
Drug: Biktarvy — Fixed dose combination preparation containing bictegravir, tenofovir alafenamide and emtricitabine
  Arms: Bictarvy

SUMMARY:
Combined antiretroviral therapy (cART) is thought to promote coronary artery disease via a number of mechanisms: abnormal lipid profiles, endothelial dysfunction, hypertension, insulin resistance and renal impairment are the main pathological mechanisms driving atherosclerosis as a consequence of cART. An association between protease inhibitors and increased cardiovascular disease risk has been shown in many large cohort trials.

CT Coronary Angiography (CTCA) is now widely used to assess for the presence of atherosclerosis, typically in patients presenting with chest pain. This imaging technique allows visualisation of the coronary arteries and quantification of any atherosclerotic disease that may be present. This technique is being increasingly used as a surrogate for cardiovascular disease risk.

HART CT is an open label, prospective, randomised-control pilot study to investigate the feasibility of performing a future appropriately powered multi-centred randomised control trial using CT based outcome data as a surrogate for cardiovascular disease risk.

Participants will be randomised to either continue their usual cART or switch to Biktarvy (a fixed dose combination of bictegravir, emtricitabine and tenofovir alafenamide). A baseline CT scan will be performed. If there is any evidence of atherosclerosis a further CT scan will be performed at the end of the study (approximately 48 weeks). This will allow quantification of any change in coronary artery plaque burden or characteristic. Participants will be also followed up for any changes in metabolic health.

ELIGIBILITY:
* HIV positive
* Undetectable viral load on cART which contain protease inhibitors (duration >6 months at eligibility visit)
* Age>40 years
* Stable cART
* No previous documented cardiovascular disease
* No contraindication to study drug
* Ability to give informed consent
* Willingness to comply with all study requirements
* No symptoms of overt cardiovascular disease

A definition of stable cART is no change to the medication regime in the preceding 6 months.

Well controlled hypertension is considered acceptable for recruitment.

Exclusion Criteria:

* Active liver disease (previously diagnosed)
* Renal disease eGFR <30
* Any ongoing infection
* Significant ionising radiation in preceding 12 months
* Known or suspected cardiovascular disease
* High dose statin therapy (Atorvastatin 20mg or more, Rosuvastatin 20mg or more)
* Pregnancy or planned pregnancy
* Breast feeding
* Allergy to iodine based contrast agent
* Known drug resistance to NRTI or Integrase
* Any contraindication to BIC/FTC/TAF
* Current enrolment onto another CTIMP.

Significant ionising radiation should not exceed >25mSv from medical sources. A definition of cardiovascular disease includes documented angina, previous myocardial infarction or previous coronary revascularization.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-03-29 (Estimated); Study Completion 2021-03-29 (Estimated)

PRIMARY OUTCOMES:
The rate of recruitment to the HART CT study | 2 years
  Rate of recruitment to the main study expressed as a rate of eligible patients screened to those who undergo randomisation.
Drop out rate | 2 years
  Drop out rate of the main study. The number of participants not completing the study expressed as a percentage of those recruited.
Change in total plaque volume (mm3) including the following derivatives: total non-calcified plaque volume (mm3), calcium volume (mm3). These derivatives will be combined to give a total plaque volume (mm3). | 2 years
  CT based quantification of coronary artery disease burden. Assessed using summary statistics and parametric or non-parametric measures of significance.
Change in Agatston Score (Agatston units). | 2 years
  Agatston calcium scoring is a highly reproducible well validated scale outlining the burden of calcific coronary artery disease. Agatston score is a function of calcium volume and density. The volume is calculated in mm3 and multiplied by a density weighting factor depending on the haunsfied units.
  Change in Agatston scores will be assessed using summary statistics and parametric or non-parametric measures of significance.
Change in segmental stenosis score | 2 years
  Coronary segments are graded as normal (no stenosis), stenosis 1%-29%, 30%-49%, 50%-69%, ≥70% by visual semiquantification method, with assignment of scores of 0, 1, 2, 3, or 4, respectively. Stenosis is not measured when the vessel diameter was <2 mm. Total segment stenosis score (TSS) per person is calculated by summing all the 15 individual SSSs with a possible score ranging from 0 to 60.
  Change in segmental stenosis scores will be assessed using summary statistics and parametric or non-parametric measures of significance.
Number of adverse plaque features | 2 years
  The change in the number of coronary segments displaying an adverse plaque characterisitc. This is defined as any one of the following (low attenuation plaque (<30 hounsfield units), positive remodelling (remodelling index >1.1), spotty calcification or napkin ring sign).
  Change in number of adverse plaque features will be assessed using summary statistics and parametric or non-parametric measures of significance.

SECONDARY OUTCOMES:
Inter and intraobserver variability of CT based outcome measures | 2 years
  To assess the inter and intraobserver variability of total plaque volume (mm3). This will be assessed for the first 20 vessels containing evidence of coronary artery disease between the two study reporters.
  The mean difference (%) will be reported.
The incidence of subclinical cardiovascular disease in the study population | 2 years
  Expressed as percentage of recruited patients.
The change in in 10-year cardiovascular disease risk between the control group and intervention group using both prediction models. | 2 years
  Summary statistics (mean) assessment of the change in 10 year cardiovascular disease risk as assessed by QRISK and ASTROCHARM risk prediction models. The 10 year cardiovascular risk will be reported as %.
  The intervention group and control group compared using parametric or non-parametric measures of significance.
Change in total cholesterol (mmol/L) including the derivatives (which are combined to give the total cholesterol) high-density lipoprotein (mmol/L), low-density lipoprotein (mmol/L) and non-high-density lipoprotein (mmol/L). | 2 years
  Intervention group and control group compared using parametric or non-parametric measures of significance. The range of cholesterol is 0-20 mmol/L
Fibroscore (Kilopascals) | 2 years
  Change from baseline to end fibroscan score. Intervention group and control group compared using parametric or non-parametric measures of significance.
  The range of KPa is 0-75.
Change in HBA1C (mmol/mol) | 2 years
  Intervention group and control group compared using parametric or non-parametric measures of significance.
  The range of HBA1C is 0-150mmol/mol.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Liverpool University Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided